CLINICAL TRIAL: NCT04195841
Title: Influence of Z Shaped Incisions on Healing and Interproximal Bone Loss in Comparison With Conventional Sulcular Incisions (H Shaped) in Implant Surgery Under Magnification: A Randomized Clinical Trial
Brief Title: Influence of Z Shaped and Conventional Sulcular Incisions on Healing and Interproximal Bone Loss in Implant Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02_D012_91553
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Bone Loss; Healing Surgical Wounds
Keywords: implant incisions; bone loss; Z shaped incision
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Two groups were made one test and control. All the subjects required rehabilitation with implants.In the test group Z shaped incision was placed. in control group sulcular H shaped incision was placed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Two horizontal incisions placed 1-2 mm away from the papilla of the teeth adjacent to the edentulous space following the mesial and distal contour of the teeth. These two horizontal incisions are then connected by an oblique incision from the disto-buccal to mesio lingual point angles.
  Interventions: Procedure: Z shaped incision
- Control group (Experimental): Sulcular incisions placed in the proximal sides of the adjacent tooth facing the edentulous space in a bucco lingual direction extending between the proximal line angles Mid crestal incision performed in the attached mucosa of the edentulous area connecting the sulcular incisions of the adjacent teeth from the distal to mesial tooth
  Interventions: Procedure: H shaped incision

INTERVENTIONS:
Procedure: Z shaped incision — After local anaesthesia, a mucoperiosteal flap will be elevated at the edentulous ridge with two horizontal incisions placed with a no MB 69 blade, 1-2 mm away from the papilla of the teeth adjacent to the edentulous space following the mesial and distal contour of the teeth. The extend of the incisions should be up to the proximal line angles of the adjacent teeth. These two horizontal incisions are then connected by an oblique incision from the disto-buccal to mesio lingual point angles. A periosteal elevator is used to elevate a full thickness mucoperiosteal flap buccally and lingually to the level of the mucogingival junction, exposing the alveolar ridge of the implant surgical sites.
  Endosseous implant placement is done followed by simple interrupted resorbable sutures
  Arms: Test group
Procedure: H shaped incision — After local anaesthesia, a mucoperiosteal flap is elelevated by placing sulcular incisions placed in the proximal sides of the adjacent tooth facing the edentulous space in a bucco lingual direction extending between the proximal line angles using a MB 69 blade.
  Mid crestal incision performed in the attached mucosa of the edentulous area connecting the sulcular incisions of the adjacent teeth from the distal to mesial tooth. A full thickness mucoperiosteal flap will be elevated buccally and lingually to the level of the mucogingival junction to expose the alveolar ridge of the implant surgical sites using a periosteal elevator.
  Endosseous implant will be placed, followed by simple interrupted resorbable sutures.
  Arms: Control group

SUMMARY:
The present study is a human, prospective, parallel, randomised controlled clinical trial conducted to check the interproximal bone loss of Z shaped incision over conventional sulcular H shaped incision.The trial is in accordance with the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.

DETAILED DESCRIPTION:
Twenty healthy individuals satisfying the inclusion and exclusion criteria were recruited for the study. A detailed, thorough medical and dental history was obtained and each patient was subjected to comprehensive clinical and radiological examination. All patients were informed about the nature of the study, the surgical procedure involved, potential benefits and risks associated with the surgical procedure and written informed consent were obtained from all patients. In the test group patients Z shaped incision was done to place implants and H shaped sulcular incision was placed in control group.

The clinical and radiographic parameters were recorded at baseline,24 hours,7days, three months and six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with single or multiple edentulous spaces in the maxillary and mandibular arches having Siebert's Class 1 and 2 ridge defects.
2. Patients willing to participate in the study.
3. Patients above 18 years of age.
4. Patients exhibiting keratinized tissue width more than or equal to 2 mm.
5. Systemically healthy patients.
6. Patients who demonstrate full mouth plaque control and bleeding scores<25% and showing good compliance.

Exclusion Criteria:

1. Patients who do not give consent.
2. Untreated periodontal disease, caries.
3. Insufficient oral hygiene.
4. Smokers.
5. Previous radiation therapy.
6. Patients with known systemic diseases and conditions
7. Pregnant and lactating women.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Inter proximal bone level | 6 months
  Mesial and distal peri-implant radiographic bone level will be recorded in millimetres on the digital radiographs with grid at baseline and follow up
Healing | 7 days
  Early wound healing index is assessed. values 1-5 is present. Increase in score depicts worse healing.

SECONDARY OUTCOMES:
Visual Analouge Score | 7 days
  a questionnaire will be given to the patients in which their responses for Visual Analog Score that ranges from 1-10 values and highest values indicate the worst outcome, variation in feeding habits, analgesics dosage is recorded.
Clinical attachment level | 3 months
  The amount of attached gingiva was measured by subtracting the probing depth from the amount of keratinised mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shobith S Mampuzha, MDS, Principal Investigator — Rajiv Gandhi University of Health Sciences; Dr Prabhuji MLV, MDS, Principal Investigator — Rajiv Gandhi University of Health Sciences
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India